CLINICAL TRIAL: NCT03611296
Title: Translational Investigation of Growth and Everyday Routines in Kids (TIGER Kids) Fitness Ancillary
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, S. Nicole Fearnbach, Assistant Professor - Research, Pennington Biomedical Research Center
Other Study IDs: 2017-009; 5T32DK064584-15 (NIH)
Record Dates: First submitted 2018-07-02; First posted 2018-08-02 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Childhood Obesity
Keywords: Cardiorespiratory fitness; Inhibitory control; Motivation; Food intake; Body composition
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Per the TIGER Kids primary study protocol, an aliquot of sample will be stored in case further tests are needed and if further consent is obtained from the subject. However, no additional samples are retained for the ancillary study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this ancillary study is to examine cardiorespiratory fitness, cognitive factors related to appetite, and objectively-measured food intake in a subsample of children and adolescents with overweight to severe obesity enrolled in the TIGER Kids prospective cohort. The primary study also collects data on habitual physical and sedentary activity, body weight and body composition, and cardiometabolic health markers.

DETAILED DESCRIPTION:
The investigators will enroll 30 boys and girls (50% female) between the ages of 10-16 years and above the 85th BMI percentile (i.e., overweight to severe obesity) in this pilot ancillary study. The objective is to examine interactions between the following energy-balance related factors:

1. Ad libitum post-exercise food intake
2. Cognitive factors, including inhibitory control, food wanting, and motivation for food
3. Exercise-related factors, including cardiorespiratory fitness, substrate utilization (carbohydrate versus fat), and perceived exertion
4. Habitual physical and sedentary activity
5. Body composition and cardiometabolic health

The prospective, longitudinal nature of the study will allow the investigators to examine these variables cross-sectionally and quantify change over two years. Of particular interest is whether cognitive factors related to energy balance, including perceived exertion, inhibitory control, food wanting, and food motivation, vary across time or are relatively stable. Finally, the investigators will assess the ability of these factors to predict changes in body composition and cardiometabolic health over two years.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for the TIGER Kids primary study
* BMI >/= 85th percentile
* Height >/= 4 feet 6 inches
* Weight < 350 pounds

Exclusion Criteria:

* Anemia
* American College of Sports Medicine (ACSM) contraindications to exercise testing (i.e., medical history of cardiovascular or pulmonary conditions, physical conditions that affect the ability to exercise)

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will identify and recruit 30 participants from the TIGER Kids primary study sample of 340 participants. Ancillary participants will be between the ages of 10-16 years and above the 85th age- and sex-specific BMI percentile (i.e., overweight to severe obesity). We will have an even distribution of boys (n=15) and girls (n=15) and aim to have a representative distribution of race.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Baseline cardiorespiratory fitness | Year 0
  Cardiorespiratory fitness, or VO2peak in mL/kg/min, is measured using a graded cycle ergometer test to volitional fatigue.
Change in cardiorespiratory fitness over 2 years | Year 0 and Year 2
  Cardiorespiratory fitness, or VO2peak in mL/kg/min, is measured using a graded cycle ergometer test to volitional fatigue.
Baseline energy intake | Year 0
  Ad libitum energy intake in kilocalories is measured using a in-laboratory dinner test-meal. Participants can eat as much or as little as they would like from the available food, which is provided in excess of energy needs.
Change in energy intake over 2 years | Year 0 and Year 2
  Ad libitum energy intake in kilocalories is measured using a in-laboratory dinner test-meal. Participants can eat as much or as little as they would like from the available food, which is provided in excess of energy needs.

SECONDARY OUTCOMES:
Baseline inhibitory control | Year 0
  Inhibitory control is measured using a Go/No-go behavioral task administered on a computer. Errors, false alarms, and reaction times are collected for various conditions: baseline, food rewards (favorite snack and least favorite snack from a selected list of options) and neutral control (unrewarded).
Change in inhibitory control over 2 years | Year 0 and Year 2
  Inhibitory control is measured using a Go/No-go behavioral task administered on a computer. Errors, false alarms, and reaction times are collected for various conditions: baseline, food rewards (favorite snack and least favorite snack from a selected list of options) and neutral control (unrewarded).
Baseline Three Factor Eating Questionnaire - Revised 18-item version 2 (TFEQ-R18v2) | Year 0
  The Three Factor Eating Questionnaire - Revised 18-item version 2 (TFEQ-R18v2) consists of three appetite-related subscales: Cognitive Restraint, Emotional Eating, and Uncontrolled Eating. Subscales are scored on a range from 0-100, with higher scores representing higher levels of that construct.
Change in Three Factor Eating Questionnaire - Revised 18-item version 2 (TFEQ-R18v2) over 2 years | Year 0 and Year 2
  The Three Factor Eating Questionnaire - Revised 18-item version 2 (TFEQ-R18v2) consists of three appetite-related subscales: Cognitive Restraint, Emotional Eating, and Uncontrolled Eating. Subscales are scored on a range from 0-100, with higher scores representing higher levels of that construct.
Baseline appetite-related Visual Analog Scales (VAS) | Year 0
  The following constructs are measured before and after the fitness test and before and after the dinner test-meal: Hunger, fullness, desire to eat, prospective food consumption, satisfaction, and wanting for specific foods (age-appropriate and commonly consumed foods for this population). VAS scores range from 0-100, with higher scores representing higher levels of that construct.
Change in appetite-related Visual Analog Scales (VAS) over 2 years | Year 0 and Year 2
  The following constructs are measured before and after the fitness test and before and after the dinner test-meal: Hunger, fullness, desire to eat, prospective food consumption, satisfaction, and wanting for specific foods (age-appropriate and commonly consumed foods for this population). VAS scores range from 0-100, with higher scores representing higher levels of that construct.

OTHER OUTCOMES:
Baseline body composition | Year 0
  In the TIGER Kids primary study, body composition is measured using whole-body dual-energy x-ray absorptiometry (DXA).
Change in body composition over 2 years | Year 0 and Year 2
  In the TIGER Kids primary study, body composition is measured using whole-body dual-energy x-ray absorptiometry (DXA).
Baseline activity patterns | Year 0
  In the TIGER Kids primary study, activity is measured for 24 hours per day over 7 consecutive days, including 2 weekend days, using ActiGraph GT3X+ accelerometers worn on the left mid-axillary line.
Change in activity patterns over 2 years | Year 0 and Year 2
  In the TIGER Kids primary study, activity is measured for 24 hours per day over 7 consecutive days, including 2 weekend days, using ActiGraph GT3X+ accelerometers worn on the left mid-axillary line.

CONTACTS AND LOCATIONS:
Overall Officials: S. Nicole Fearnbach, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fearnbach SN, Johannsen NM, Martin CK, Katzmarzyk PT, Beyl RA, Hsia DS, Carmichael OT, Staiano AE. A Pilot Study of Cardiorespiratory Fitness, Adiposity, and Cardiometabolic Health in Youth With Overweight and Obesity. Pediatr Exerc Sci. 2020 Apr 25;32(3):124-131. doi: 10.1123/pes.2019-0192. PMID 32335525
- [Background] Fearnbach N, Staiano AE, Johannsen NM, Hsia DS, Beyl RA, Carmichael OT, Martin CK. Predictors of Post-Exercise Energy Intake in Adolescents Ranging in Weight Status from Overweight to Severe Obesity. Nutrients. 2022 Jan 5;14(1):223. doi: 10.3390/nu14010223. PMID 35011098